CLINICAL TRIAL: NCT05487872
Title: Mindfulness Skills Training and Psychological Inflexibility: a Randomized Trial
Brief Title: Mindfulness and Psychological Inflexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahcesehir Cyprus University (Other)
Responsible Party: Principal Investigator, Buse Keskindag, Principal Investigator, Bahcesehir Cyprus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BAU/EK-2022/02
Record Dates: First submitted 2022-07-30; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Mindfulness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audio-guided mindfulness skills training (Other): Participants in this group listened to a 15 mins audio track to practice mindfulness exercises
  Interventions: Behavioral: Mindfulness skills training to reduce experiential avoidance and anxiety symptoms
- Virtual reality (VR) -based mindfulness skills training (Experimental): Participants in this group completed mindfulness exercises on the VR system. The system included the same 15 mins audio track and additionally a video that displayed a 360° spherical landscape view of the sea in the afternoon
  Interventions: Behavioral: Mindfulness skills training to reduce experiential avoidance and anxiety symptoms

INTERVENTIONS:
Behavioral: Mindfulness skills training to reduce experiential avoidance and anxiety symptoms — The intervention aimed to increase participants' mindfulness skills which may be critical in decreasing general experiential avoidance and anxiety symptoms

SUMMARY:
This study aimed to examine whether mindfulness skills training can help to reduce experiential avoidance and anxiety level. This study investigated whether the training delivery methods (audio-guided mindfulness exercise or virtual reality-based mindfulness exercise) differ in terms of changing general experiential avoidance and anxiety symptoms.

DETAILED DESCRIPTION:
The experimental design (randomized trial) was used in this study. Data were collected through convenience sampling. After obtaining ethical approval fromEthics Committee of the Bahçeşehir Cyprus University, participants were invited to participate in the study via advertisements posted in the university building. Recruited participants were randomly assigned to the experimental group or control group. All participants will be provided with an informed consent form which provided information about participant's right and data management. Participants in the experimental group completed mindfulness exercise on Virtual Reality (VR) system where they listened to an audio track (guide for the exercise) and saw calming nature scenes (e.g., views on the beach) whereas those in the control group completed mindfulness exercise by listening to the (same) audio track only. Each mindfulness session took approximately 15 mins. In total, four sessions were completed in two weeks (2 sessions per week). After obtaining informed consent, the participants completed a survey pack that included valid and reliable measurement scales (mindfulness skills [The Cognitive and Affective Mindfulness Scale - Revised], experiential avoidance [Acceptance and Action Questionnaire-II], and anxiety symptoms [Generalized Anxiety Disorder Scale]) at two-time points (i.e., pre-test [before intervention], and post-test [after 4 sessions/when sessions were completed], At the end of the study, the participants were provided with a debrief form.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 and above,
* ability to read, and/or understand English

Exclusion Criteria:

* Participants who regularly practice mindfulness exercise were excluded form the analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Change in experiential avoidance | at two time points (pre-intervention and immediately after the intervention)
  Experiential avoidance is an example of psychological inflexibility. Experiential avoidance was measured via Acceptance and Action Questionnaire-II. The scale includes 7 items that are rated on a seven-point scale (1 = never true - 7 = always true). The minimum and maximum scores on the scale range between 7 and 49 points. Higher scores on the scale indicate greater experiential avoidance (psychological inflexibility)

SECONDARY OUTCOMES:
Change in anxiety | at two time points (pre-intervention and immediately after the intervention)
  Anxiety symptoms were measured via Generalized Anxiety Disorder Scale. The scale includes 7 items rated on 4 point scale (0 = Not at all, 1 = Several days, 2 = More than half of the days - 3 = Nearly every day). Scores 5, 10, 15 obtained from the test indicate mild, moderate, and severe anxiety, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Buse Keskindag, Principal Investigator — Bahcesehir Cyprus University
Locations (1):
- Bahçeşehir Cyprus University, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No